CLINICAL TRIAL: NCT03504514
Title: Evaluation of the Effect of a Speech Detection Tool on the Improvement of Phonation in Neuromuscular Patients Dependent on Mechanical Ventilation
Acronym: Ventiphono
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-A00109-44
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-08

CONDITIONS: Neuromuscular Diseases; Mechanical Ventilation; Speech
Keywords: non invasive ventilation; invasive ventilation; neuromuscular disorder; phonation; speech
MeSH Terms: conditions — Neuromuscular Diseases; Speech

STUDY DESIGN:
Intervention Model Description: monocentric, open, randomized, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional mechanical ventilation (No Intervention): Conventional mechanical ventilation, with patient ventilator usual parameters
- Adapted mechanical ventilation (Experimental): Mechanical ventilation with parameters specifically modified to improve speech the effect is evaluated with speech trials during different ventilation conditions
  Interventions: Device: speech trials during different ventilation conditions; Other: speech trial

INTERVENTIONS:
Device: speech trials during different ventilation conditions — ventilator parameters are modified
  Arms: Adapted mechanical ventilation
Other: speech trial — reading duration, vocal flow, intelligibility and voice quality will be evaluated during speech
  Arms: Adapted mechanical ventilation

SUMMARY:
Ventilation is a major treatment of respiratory failure due to neuromuscular disorders. First line treatment is noninvasive ventilation (NIV) but in some situations, especially in case of NIV inefficiency, invasive ventilation with tracheostomy (IVT) may be required. In both situations, patients may become dependent on ventilatory support with the disease evolution. Ventilation then can interfere speech and the quality of communication of the patients. Modification of the ventilation parameters may result in improved speech quality (for example, positive expiratory pressure (PEP) while not necessary for ventilation quality can dramatically improve speech in tracheostomized patients). Therefore, it would be of interest to allow patients to benefit from these specific parameters when they need to speak without maintaining them when patients are not speaking. We want to evaluate a specific ventilator feature which can detect speech and switch to specific ventilation parameters adapted for speech We believe that this feature will improve significantly speech quality in patients dependant either on NIV or IVT.

DETAILED DESCRIPTION:
Nowadays, the first line treatment of chronic respiratory failure in neuromuscular disorder is non invasive ventilation (NIV). However, while NIV can compensate the respiratory disability and significantly delays significantly the necessity for invasive ventilation with a tracheostomy (IVT), it is used for significant periods of time during daytime in patients with severe respiratory failure and can therefore interfere with patients' speech. Moreover, if NIV becomes inefficient, IVT may be required to pursue ventilatory support to treat the respiratory failure; tracheostomy also interferes with phonation and specific adaptations are necessary to optimize phonation and speech quality.

Adaptation of ventilation parameters (mainly triggering sensitivity and use of positive expiratory pressure (PEP)) can significantly improve speech quality and therefore ventilated patients' communication. These adapted parameters are not strictly necessary for ventilation outside of speaking periods. It would be of interest to be able to use them exclusively during speech. In neuromuscular patients, the major motor disability constitutes a challenge as most patients are unable to use themselves the controls of their ventilator (and to potentially switch to a speech adapted ventilation program). We want to evaluate a device able to automatically detect speech and to transitorily switch from the patient's usual ventilation parameters to speech specific parameters set to optimize phonation quality.

Specific adaptations differs between NIV or IVT, therefore we will evaluation two groups of ventilation dependent patients divided according to their ventilation mode.

We believe that this device may improve the speech of NIV patients as well as IVT patients. Patients would benefit from an appropriate ventilator support without any ventilation desynchronization during speech. Speech would be more fluent and natural which would result in improved communication.

Objectives The main objective of this study is to demonstrate that phonation is improved by the use of a device allowing the transitory switch to specific speech parameters of ventilation in neuromuscular ventilator dependent patient whether during NIV or during IMT.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age > or equal to 18)
* Neuromuscular patients with a restrictive respiratory failure without major bulbar involvement.
* Adult patient.
* Ventilator dependancy= ventilation duration of 16h/day or more either with NIV or IMT
* Leak ventilation for IMT patients
* Respiratory autonomy of at leat 1h per day
* Usual ventilation mode : assist control mode (either pressure or volume controlled mode) ou spontaneous breathing mode with target volume
* Stable hemodynamic state
* Signed informed consent

Exclusion Criteria:

* Refusal to participate
* Use of cuffed tracheostomy tube
* Inability to read
* Pregnancy
* Protected adults
* Acute respiratory failure
* Hemodynamic instability
* not registered with the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
reading duration | 15 minutes
  duration for reading a specific text in seconds

SECONDARY OUTCOMES:
Vocal flow | 15 minutes
  vocal flow in syllables/second during the reading of a specific text
vocal range | 2 minutes
  vocal range from lowest to highest pitch
intelligibility | 15 minutes
  evaluation of intelligibility during reading evaluated by listeners blinded to ventilation conditions
Speech quality | 5 min
  evaluation of prosodia by listeners blinded to ventilation conditions
Speech quality | 1 minute
  evaluation of speech quality by the patient using a visual analogical scale
Speech comfort | 1 minute
  evaluation of speech comfort by the patient using a visual analogical scale
Respiratory comfort | 1 minute
  evaluation of respiratory comfort by the patient using a visual analogical scale
dyspnea | 1 minute
  evaluation of dyspnea during speech evaluated with the modified Borg scale (ranking from 0 to10)
oxygen saturation | 15 min
  evaluation of Respiratory tolerance during speech by measuring oxygen saturation
respiratory rate | 15 min
  evaluation of Respiratory tolerance during speech by measuring respiratory rate
cardiac frequency | 15 min
  evaluation of Cardiovascular tolerance during speech by measuring cardiac frequency
Patient satisfaction | 1 minute
  evaluation of Patient satisfaction with speech with the ventilation mode by the patient using a visual analogical scale

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Prigent, MD PhD, Principal Investigator — Raymond Poincaré Hospital
Locations (1):
- Raymond Poincaré hospital, Garches, France

IPD SHARING:
Plan to Share IPD: No